CLINICAL TRIAL: NCT01615276
Title: The Effect of Neuromuscular Electrical Stimulation on Post-prandial Muscle Protein Accretion in Healthy Elderly Men
Brief Title: Neuromuscular Electrical Stimulation (NMES) and Muscle Protein Accretion (ES-PRO)
Acronym: ES-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MEC 12-3-020
Record Dates: First submitted 2012-05-30; First posted 2012-06-08 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Sarcopenia
Keywords: Neuromuscular Electrical Stimulation; Ageing; Protein ingestion
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein ingestion (Placebo Comparator): Protein ingestion directly after the contralateral leg received NMES
  Interventions: Device: No Enraf Nonius Tensmed S84 for Neuromuscular electrical stimulation (NMES) NMES
- Protein ingestion after NMES (Experimental): Ingestion of intrinsically labeled protein, directly after one hour of Neuromuscular electrical stimulation (NMES)
  Interventions: Device: Enraf Nonius Tensmed S84 for Neuromuscular electrical stimulation (NMES)

INTERVENTIONS:
Device: Enraf Nonius Tensmed S84 for Neuromuscular electrical stimulation (NMES) — One our of one-legged neuromuscular electrical stimulation (NMES)
  Arms: Protein ingestion after NMES
Device: No Enraf Nonius Tensmed S84 for Neuromuscular electrical stimulation (NMES) NMES — No neuromuscular electrical stimulation (NMES) will be applied in the control leg
  Arms: Protein ingestion

SUMMARY:
In the present study, the effect of a bolus of intrinsically labeled milk directly after one-legged NMES will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 65 - 85 years
* 18.5 < BMI < 30 kg∙m2

Exclusion Criteria:

* Type II diabetes
* All co morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthrosis, arthritis, spasticity/rigidity, all neurological disorders, paralysis, hip/knee surgery).
* Use of anticoagulants, blood diseases, allergy for lidocaine
* Use of NSAIDs and acetylsalicylic acid
* Patients suffering from PKU (Phenylketonuria)
* Presence of implantable cardioverter defibrillator and/or pacemaker
* Performed regular resistance type exercise in the past 6 months

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Tracer enrichment in the muscle biopsy | 4 hours after protein ingestion

SECONDARY OUTCOMES:
Fractional synthetic rate (FSR) | 0-4 hours after protein ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356